CLINICAL TRIAL: NCT03202927
Title: A Randomized, Single Blind, Repeat-dose, Two Cycle, Parallel-Arm Comparative Immunogenicity Study Comparing TPI-120 to Neulasta® in Healthy Adult Subjects
Brief Title: Comparative Immunogenicity Study Comparing TPI-120 to Neulasta® in Healthy Adult Subjects
Acronym: TPI-120
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adello Biologics, LLC (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Principal Investigator, Dr. Prayag Shah, principal investigator, Adello Biologics, LLC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADL-CL-112
Record Dates: First submitted 2017-04-25; First posted 2017-06-29 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — pegfilgrastim

STUDY DESIGN:
Intervention Model Description: This is a single blind parallel comparative immunogenicity study
Who Masked: Participant
Masking Description: As this is single blind study so study participants would be blinded in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TPI-120 (PEGFILGRASTIM) (Experimental): One daily dose of TPI-120 (PEGFILGRASTIM) 6 mg/0.6 ml administered subcutaneously on Day 1 (Study Day 1) of Cycle 1 followed by one daily dose of 6 mg/0.6 ml administered subcutaneously on Day 1 (Study Day 22) of Cycle 2 with a gap of 21 days between two cycles
  Interventions: Drug: PEGFILGRASTIM
- Neulasta (PEGFILGRASTIM) (Active Comparator): One daily dose of Neulasta (PEGFILGRASTIM) 6 mg/0.6 ml administered subcutaneously on Day 1 (Study Day 1) of Cycle 1 followed by one daily dose of 6 mg/0.6 ml administered subcutaneously on Day 1 (Study Day 22) of Cycle 2 with a gap of 21 days between two cycles
  Interventions: Drug: PEGFILGRASTIM

INTERVENTIONS:
Drug: PEGFILGRASTIM — Pegfilgrastim is a covalent conjugate of recombinant methionyl human granulocyte colony-stimulating factor and monomethoxy polyethylene glycol.
  Other Names: PEG GCSF, Neulasta

SUMMARY:
This study will compare treatment emergent incidence rate of ADA between TPI-120 and US licensed Neulasta in normal healthy adult subjects

DETAILED DESCRIPTION:
Healthy subjects have been selected as the study population for this comparative study because this population is more homogenous with respect to immune response and offers significant advantages with regards to recruitment and logistical aspects. This study will comprise of two cycles with each cycles will have a single dose of PEG FILGRASTIM administration to all study subjects as per the randomization schedule. Subjects will be confined from at least 10 hours prior to dosing, at the time indicated by the CRU, until 36 hours post-dose on day 2 in each Cycle. Dosing in each Cycle are separated by 21 days.

Subjects will return for all subsequent blood draws and ADA assessments, as indicated in The Schedule of Event

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, non-smoker (no use of tobacco or nicotine products within 3 months prior to dosing), 19 - 55 years of age (inclusive), with body mass index (BMI) ≥ 19 and ≤ 30 kg/m2, and body weight not < 50 kg or > 100 kg at the time of screening.
2. Healthy as defined by:

   1. The absence of clinically significant (in the opinion of the PI/designee) illness or surgery within 4 weeks prior to initial dosing.
   2. The absence of a clinically significant (in the opinion of the PI/designee) history of disease.
   3. WBC (white blood cell) > 4.0 x 109/L and < 1.5 times the upper limit of normal (ULN), ANC (absolute neutrophil count) > 2.0 x 109/L and < 1.5 times the upper limit of normal (ULN), Platelet count > 150 x 109/L, AST (aspartate aminotransferase) < 2.5 time the upper limit of normal (ULN), ALT (alanine aminotransferase) < 2.5 time the upper limit of normal (ULN), Serum bilirubin < 1.5 time the upper limit of normal (ULN) and Serum creatinine < 1.5 time the upper limit of normal (ULN) at the time of screening. [Refer to APPENDIX 1 for normal reference ranges]
   4. The absence of febrile (defined by a documented oral temperature of 101.5 °F or greater) or infectious illness within 1 week of first dosing.
   5. The absence of a clinically significant history of skin disorders, including psoriasis.
3. Females of childbearing potential must be willing to use acceptable contraceptive methods throughout the study, and for 30 days thereafter.
4. Females of non-childbearing potential must have undergone sterilization procedures, at least 6 months prior to the first dose or be postmenopausal with amenorrhea for at least 1 year prior to the first dose and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status
5. Capable and willing of consent.
6. Male subjects willing to follow approved birth control method for the duration of the study, and for 30 days thereafter, such as (a double barrier method) condom with spermicide, condom with diaphragm or abstinence, subject should also not donate sperm during this time.

Exclusion Criteria:

1. Any positive test for hepatitis B, hepatitis C, or HIV at the time of screening.
2. Illicit/illegal drug use as evidenced by a positive drug screen at screening or check -in.
3. Positive result for urine alcohol test at screening or check-in
4. Tobacco use as evidenced by a positive cotinine result at screening or check-in.
5. History of allergic reactions to pegfilgrastim, filgrastim, Escherichia coli (E. coli)-derived proteins, or other related drugs. History of allergic reactions or hypersensitivity to acetate/acetic acid, polysorbate 20, or sorbitol.
6. Hereditary fructose intolerance.
7. Females with positive pregnancy tests at screening or check-in.
8. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study or completing follow-up activities.
9. Clinically significant ECG or vital signs abnormalities at screening.
10. History of significant alcohol abuse within one year prior to initial dosing or regular use of alcohol (more than 14 units of alcohol per week) within six months prior to initial dosing.
11. History of drug abuse or use of illicit/illegal drugs within 1 year prior to initial dosing.
12. No medications are permitted during the study. Exceptions are:

    1. Hormonal contraceptives and Hormone Replacement Therapy (HRT),
    2. Thyroid replacement therapy i.e., liothyronine (T3) or levothyroxine (T4).
    3. Acetaminophen
13. Donation of plasma within 7 days of initial dosing; blood donation or significant loss of blood within 30 days of initial dosing.
14. Participation in a clinical trial involving the administration of an investigational drug or marketed drug within 30 days prior to initial dosing (90 days for biologics) or concomitant participation in an investigational study involving no drug administration.
15. Females who are breast-feeding or lactating.
16. History of pulmonary infiltrate or pneumonia (radiologically confirmed) within 6 months prior to initial dosing.
17. Any past exposure to recombinant human G-CSF products and/or a known history of prior treatment with blood-cell colony stimulating factors, interleukins or interferons.
18. History of cancer
19. Subjects who are on a special diet or who have self-reported a weight loss of more than 15 pounds within 1 month prior to initial dosing.
20. Acute viral or bacterial infection within 1 month prior to initial dosing only if considered clinically significant in the opinion of the Principal Investigator/designee.
21. History of any clinically significant disease or condition that, in the opinion of the Principal Investigator/designee, would render them unsuitable for inclusion in the study.
22. Any vaccination (including influenza) within 90 days prior to initial dosing.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2017-03-25 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Treatment emergent ADA incidence rate | Pre dose Day 1 (Day 1 of Cycle 1), Day 8 ± 1, Day 21 ± 1, prior to dosing on Day 1 of Cycle 2), Day 29 ± 1, Day 58 ± 1
  Treatment emergent ADA levels for TPI-120 and Neulasta® will be estimated and compared to evaluate potential differences between the two products in the incidence of ADA human immune responses

SECONDARY OUTCOMES:
Safety Variable - Tolerability as measured by Injection Site reactions | 0.5, 2, 4, 6, 12 (Day 1), 24 (Day 2) hours post dose in each cycle
  Tolerability as measured by Injection Site reactions
Safety Variable - Immunogenicity as measured by presence of Anti Drug Antibodies | Day 1 of Cycle 1, On Study Day 8 ± 1, On Study Day 21 ± 1, Day 1 of Cycle 2), On Study Day 29 ± 1, On Study Day 58 ± 1
  Immunogenicity as measured by presence of Anti Drug Antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Cui, MD, Study Director — Adello Biologics, LLC
Locations (2):
- United States (2):
  - Celerion Inc., Tempe, Arizona
  - Celerion Inc., Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: No
Sponsor will decide later on